CLINICAL TRIAL: NCT02748798
Title: Developing Optimal Parameters for Hyperpolarized Noble Gas (3He and 129Xe) and Inert Fluorinated Gas Magnetic Resonance Imaging of Lung Disorders
Brief Title: Developing Optimal Parameters for Hyperpolarized Noble Gas and Inert Fluorinated Gas MRI of Lung Disorders
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding is no longer available due to the failure to enroll the target number of participants within the required timeframe.
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Collaborators: Thunder Bay Regional Health Sciences Centre (Other); St. Joseph's Care Group (Other); Lakehead University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RP-312-07112014
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Transplant; Lung Resection; Lung Cancer; Asthma; Cystic Fibrosis; Chronic Obstructive Pulmonary Disease; Emphysema; Mesothelioma; Asbestosis; Pulmonary Embolism; Interstitial Lung Disease; Pulmonary Fibrosis; Bronchiectasis; Seasonal Allergies; Cold Virus; Lung Infection; Pulmonary Hypertension; Pulmonary Dysplasia; Obstructive Sleep Apnea
MeSH Terms: conditions — Lung Neoplasms; Asthma; Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive; Emphysema; Mesothelioma; Asbestosis; Pulmonary Embolism; Lung Diseases, Interstitial; Pulmonary Fibrosis; Bronchiectasis; Rhinitis, Allergic, Seasonal; Hypertension, Pulmonary; Sleep Apnea, Obstructive | interventions — perflutren; Sulfur Hexafluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Experimental): Participants will inhale investigational gases (HP 3He, HP 129Xe, PFP and SF6) according to the procedure for that intervention. All participants can potentially inhale all the gases. Magnetic resonance imaging will be performed during breath-holds or continuous breathing (gas-dependent) with the appropriate investigational human lung coil (3He Human Lung Coil, 129Xe Small and Large Human Lung Coil, or PFP and SF6 Human Lung Coil), using the 3T Research MRI at the Thunder Bay Regional Health Sciences Centre.
  Interventions: Drug: HP 3He; Drug: HP 129Xe; Drug: PFP; Drug: SF6; Device: 129Xe Small and Large Human Lung Coil; Device: 3He Human Lung Coil; Device: PFP and SF6 Human Lung Coil
- Lung Disorder Participants (Experimental): Participants will inhale investigational gases (HP 3He, HP 129Xe, PFP and SF6) according to the procedure for that intervention. All participants can potentially inhale all the gases. Magnetic resonance imaging will be performed during breath-holds or continuous breathing (gas-dependent) with the appropriate investigational human lung coil (3He Human Lung Coil, 129Xe Small and Large Human Lung Coil, or PFP and SF6 Human Lung Coil), using the 3T Research MRI at the Thunder Bay Regional Health Sciences Centre.
  Interventions: Drug: HP 3He; Drug: HP 129Xe; Drug: PFP; Drug: SF6; Device: 129Xe Small and Large Human Lung Coil; Device: 3He Human Lung Coil; Device: PFP and SF6 Human Lung Coil

INTERVENTIONS:
Drug: HP 3He — 3He will be hyperpolarized using a custom-built polarizer to enhance its MRI signal. Hyperpolarization does not change the chemical or physical properties of helium gas.
  Other Names: Hyperpolarized helium 3
Drug: HP 129Xe — 129Xe will be hyperpolarized using a Xemed polarizer to enhance its MRI signal. Hyperpolarization does not change the chemical or physical properties of xenon gas.
  Other Names: Hyperpolarized xenon 129
Drug: PFP — Perfluoropropane (PFP) will be premixed and delivered to the participants with no further processing.
  Other Names: Perfluoropropane
Drug: SF6 — Sulfur hexafluoride (SF6) will be premixed and delivered to the participant with no further processing.
  Other Names: Sulfur hexafluoride
Device: 129Xe Small and Large Human Lung Coil — The investigational 129Xe small and large quadrature lung coils are sensitive to 129Xe resonant frequencies and therefore will be paired with the investigational drug 129Xe. The size of the coil used will depend on the participants' body size.
Device: 3He Human Lung Coil — The investigational 3He quadrature lung coil is sensitive to 3He resonant frequencies and therefore will be paired with the investigational drug 3He.
Device: PFP and SF6 Human Lung Coil — The investigational PFP and SF6 quadrature lung coil is sensitive to inert fluorinated gas resonant frequencies and therefore will be paired with both PFP and SF6.

SUMMARY:
The goal of this research is to optimize the MRI system to obtain ideal lung images using Hyperpolarized (HP) Noble and Inert Fluorinated Gases as contrast agents. Lung coils tuned to the frequencies of these gases will be used. This study will take place at TBRHSC in the Cardiorespiratory Department and in the Research MRI facility.

DETAILED DESCRIPTION:
MR images of the lung obtained using HP 3He, HP 129Xe, and inert fluorinated gases essentially show the distribution of the inhaled gas inside the lungs. Measurements can be performed on these images to provide additional information that can be related to pulmonary function.

Participation will involve at least two study visits. During the first visit, participants will provide written, informed consent, and undergo eligibility screening. Study drug administration, use of the investigational devices, and MR imaging for this study will be performed at the 3T Research MRI at the Thunder Bay Regional Health Sciences Centre (TBRHSC). Pulmonary Function Tests (PFTs) will be performed at TBRHSC by a Registered Respiratory Therapist (RRT) and an MR Tech will be present for the duration of participant scans.

Participants will be placed in the MRI with the appropriate chest coil wrapped around them like a vest. Several inhalation procedures will be carried out during scanning. Participants safety will be closely monitored throughout the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Is either:

  1. A healthy volunteer (i.e.: someone not diagnosed with a lung disorder written below; this may include smokers who have not been diagnosed with a lung disorder) or
  2. Has been diagnosed with one of the following respiratory disorders: lung transplants, lung resection, lung cancer, asthma, cystic fibrosis, chronic obstructive pulmonary disease, emphysema, mesothelioma, asbestosis, pulmonary embolism, interstitial lung disease, pulmonary fibrosis, bronchiectasis, seasonal allergies, pneumonia, cold virus, lung infection, pulmonary hypertension, pulmonary dysplasia, obstructive sleep apnea
* Able to provide informed consent
* Able to hold their breath for imaging:

  1. Healthy volunteers enrolled in this study must be able to hold their breath for 25 seconds
  2. Lung disorder participants must be able to hold their breath for 15 seconds

Exclusion Criteria:

* Have contraindication to MR imaging (i.e. ferrous implants, cardiac pacemakers) - determined by MR screening prior to scans.
* Have a history of claustrophobia.
* Female exclusion only: are or may be pregnant.
* Requires an oxygen mask and cannot use a nasal cannula.
* Blood oxygen saturation is below 92% (measured at rest in a sitting position, and with an O2 nasal cannula if the participant normally uses one).
* Has had an acute respiratory infection in the past 10 days.
* Is a student currently enrolled in a course at Lakehead University where the Principal Investigator (PI) is the instructor.
* Is a student currently enrolled in a degree program at Lakehead University where the PI is their direct thesis supervisor.
* Is currently an employee of the PI at the Thunder Bay Regional Research Institute (TBRRI) and/or Lakehead University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-10-16 (Actual); Study Completion 2021-10-16 (Actual)

PRIMARY OUTCOMES:
Signal to Noise Ratio | 2 years
  The primary objective of this study is to determine an optimized set of scan parameters that will produce clear, anatomically and clinically relevant images of the lungs for healthy participants and various types of lung disorder participants, and using one or more gas type (3He, 129Xe, PFP, SF6).

SECONDARY OUTCOMES:
Correlation with PFTs | 2 years
  The secondary objective of this study is to correlate the results with PFTs, including spirometry and plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell S Albert, PhD, Principal Investigator — Thunder Bay Regional Health Research Institute
Locations (1):
- Thunder Bay Regional RI, Thunder Bay, Ontario, Canada

REFERENCES:
- [Background] Couch MJ, Blasiak B, Tomanek B, Ouriadov AV, Fox MS, Dowhos KM, Albert MS. Hyperpolarized and inert gas MRI: the future. Mol Imaging Biol. 2015 Apr;17(2):149-62. doi: 10.1007/s11307-014-0788-2. PMID 25228404
- [Result] Kooner HK, McIntosh MJ, Matheson AM, Venegas C, Radadia N, Ho T, Haider EA, Konyer NB, Santyr GE, Albert MS, Ouriadov A, Abdelrazek M, Kirby M, Dhaliwal I, Nicholson JM, Nair P, Svenningsen S, Parraga G. 129Xe MRI ventilation defects in ever-hospitalised and never-hospitalised people with post-acute COVID-19 syndrome. BMJ Open Respir Res. 2022 May;9(1):e001235. doi: 10.1136/bmjresp-2022-001235. PMID 35584850
- [Result] Matheson AM, McIntosh MJ, Kooner HK, Lee J, Desaigoudar V, Bier E, Driehuys B, Svenningsen S, Santyr GE, Kirby M, Albert MS, Shepelytskyi Y, Grynko V, Ouriadov A, Abdelrazek M, Dhaliwal I, Nicholson JM, Parraga G. Persistent 129Xe MRI Pulmonary and CT Vascular Abnormalities in Symptomatic Individuals with Post-acute COVID-19 Syndrome. Radiology. 2022 Nov;305(2):466-476. doi: 10.1148/radiol.220492. Epub 2022 Jun 28. PMID 35762891